CLINICAL TRIAL: NCT03589937
Title: A Longitudinal Study on Ocular Development and Refractive Error Changes Among children-and Adolescent
Brief Title: Ocular Development and Refractive Error Changes Among Children and Adolescent - A Longitudinal Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yizhi Liu, Professor, Zhongshan Ophthalmic Center, Sun Yat-sen University
Other Study IDs: SYSU-OPH-004
Record Dates: First submitted 2018-06-20; First posted 2018-07-18 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Myopia
Keywords: refractive error; ocular structural parameters
MeSH Terms: conditions — Myopia; Refractive Errors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims to observe the ocular development and refractive error changes among school children and adolescents

DETAILED DESCRIPTION:
This study aims to observe the refractive error changes of school children and adolescents for 3 years, and to collect data of ocular structural parameters, family history and environmental factors so as to understand the natural course and internal laws of myopia progression.

ELIGIBILITY:
Inclusion Criteria:

* School children and adolescent at the age of 3(Junior Kindergarten), 6(Grade 1), 9(grade 4), 12(grade 7).
* No allergy to tropicamide or topical anesthetics
* written informed consent is obtained from guardian
* Be willing to cooperate with the relevant ophthalmological examination and complete the questionnaire.

Exclusion Criteria:

* No history of eye diseases
* Receiving or has been received treatment of myopia control such as atropine eye drops, corneal contact lens or myopic glasses
* A history of allergy to topic amide or topical anesthetics
* Have severe systemic disease
* Missing ability to give informed consent

Ages: 3 Years to 12 Years | Sex: All
Age Groups: Child
Study Population: School children and adolescent at the age of 3(Junior Kindergarten), 6(Grade 1), 9(grade 4), 12(grade 7)
Sampling Method: Non-Probability Sample
Enrollment: 7050 (Actual)
Dates: Start 2018-07-20 (Actual); Primary Completion 2024-07-20 (Estimated); Study Completion 2024-07-20 (Estimated)

PRIMARY OUTCOMES:
spherical equivalent change | examine every 12 months, follow up for 3 years
  SE was measured by autorefractometer with cycloplegic once a year at scheduled time Every 12 months, follow up for 3 years

SECONDARY OUTCOMES:
Axial length | examine every 12 months, follow up for 3 years
  Axial length is measured by IOMaster once a year at scheduled time
Anterior chamber depth | examine every 12 months, follow up for 3 years
  Anterior chamber depth is measured by IOMaster once a year at scheduled time
lens thickness | examine every 12 months, follow up for 3 years
  lens thickness is measured by IOMaster once a year at scheduled time
Vitreous length | examine every 12 months, follow up for 3 years
  Vitreous length was measured by IOMaster once a year at scheduled time
Environmental factor | examine every 12 months, follow up for 3 years
  Time of outdoor activities & short range reading,measured by questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Yizhi LIU, PhD, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-san University
Locations (1):
- Zengcheng, Guangzhou, Guangdong, China